CLINICAL TRIAL: NCT05787665
Title: Evaluation of the Impact of Lung Ultrasound on Mortality and Rehospitalization in Patients Admitted to the Emergency Department With Dyspnea: a Prospective Observational Cohort
Brief Title: Evaluation of the Impact of Lung Ultrasound on Mortality and Rehospitalization in Patients Admitted to the Emergency Department With Dyspnea
Acronym: HOSPITALUS
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL23_0002; 2023-A00177-38 (Other: ANSM)
Record Dates: First submitted 2023-03-15; First posted 2023-03-28 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Dyspnea
Keywords: Lung ultrasonography; emergency department; mortality; rehospitalization
MeSH Terms: conditions — Dyspnea; Emergencies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- With Lung Ultrasonography: Patient who meet inclusions criteria, and which lung ultrasonography were performed during their medical care in Emergency Department
  Interventions: Other: phone call at 3 months
- Without Lung Ultrasonography: Patient who meet inclusions criteria, and which lung ultrasonography were not performed during their medical care in Emergency Department.
  Interventions: Other: phone call at 3 months

INTERVENTIONS:
Other: phone call at 3 months — patients will be called at 3 months to know if they are alive and to know if they have been rehospitalized

SUMMARY:
Dyspnea is a frequent reason for referral to emergency departments, leading to a 30-day mortality rate of up to 10% and a 3-month rehospitalization rate of over 30%.

Multiple etiologies, as well as poor performance of clinical examination and chest radiography, lead to a diagnostic error rate of nearly 30% at the end of emergency department care. These diagnostic errors lead to rehospitalization and an excess mortality rate of more than 50% compared to patients with a correct initial diagnosis, which is explained in particular by the use of inappropriate therapies.

Lung ultrasound is a rapid, non-irradiating, non-invasive, inexpensive, reproducible imaging test that can be used at the bedside. It has a better diagnostic performance than chest radiography, commonly performed in emergency departments.The immediate benefit of lung ultrasound for the most common diagnoses in emergency medicine has already been demonstrated.

From an organizational point of view, a few studies have shown a benefit of lung ultrasound in reducing the time spent in emergency departments and the number of additional examinations necessary for the final diagnosis. However, there is no data in the literature on the longer term impact of its use in the emergency department.

The primary objective is to evaluate the impact of performing lung ultrasound in terms of 3-month mortality and rehospitalization as part of the diagnostic process for patients admitted to the emergency department with dyspnea.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Admission to the emergency department with dyspnea defined by:

The functional sign of dyspnea experienced by the patient; Or a clinical sign of respiratory distress.

- Non-opposition of the patient or patient's family if the patient isn't able

Exclusion Criteria:

* Trauma-induced dyspnea;
* Patient being on palliative care;
* Patient with criteria for initial resuscitation with admission to a critical care unit;
* Pregnant women, women in labour or nursing mothers;
* Persons deprived of liberty by judicial or administrative decision;
* Persons under psychiatric care;
* Persons admitted to a health or social institution for purposes other than research;
* Persons of full age subject to a legal protection measure (guardianship, curatorship);

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will focus on adult patients consulting for dyspnea in the emergency department of the Edouard-Herriot Hospital (HCL).
Sampling Method: Non-Probability Sample
Enrollment: 385 (Actual)
Dates: Start 2023-06-16 (Actual); Primary Completion 2025-11-28 (Actual); Study Completion 2025-11-28 (Actual)

PRIMARY OUTCOMES:
The primary objective is to evaluate the impact of performing lung ultrasound in terms of 3-month mortality as part of the diagnostic process for patients admitted to the emergency department with dyspnea. | at 3 months
  The primary endpoint is the rate of mortality at 3 months.
The primary objective is to evaluate the impact of performing lung ultrasound in terms of 3-month rehospitalization as part of the diagnostic process for patients admitted to the emergency department with dyspnea. | at 3 months
  the primary endpoint is the rate of rehospitalization at 3 months

CONTACTS AND LOCATIONS:
Overall Officials: JULIA MORERE, MD, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Hôpital Edouard-Herriot - Emergency Department, Lyon, France